CLINICAL TRIAL: NCT01021540
Title: Prospective Study Evaluating the Effect of Repository Corticotropin in the Treatment of Various Nephrotic Syndromes
Acronym: ACTH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Arizona Kidney Disease and Hypertension Center (Other)
Responsible Party: Sungchun Lee, MD, AKDHC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009003
Record Dates: First submitted 2009-11-25; First posted 2009-11-30 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Nephrotic Syndromes
Keywords: Nephritis,Nephropathy
MeSH Terms: conditions — Nephrotic Syndrome; Nephritis; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Repository corticotrophin — Acthar 80 IU SQ once a week and titrated up to twice a week
  Other Names: H.P. Acthar Gel

SUMMARY:
To determine if H.P. Acthar Gel (repository corticotrophin) has the same anti-proteinuric effects seen with the synthetic ACTH analogue in Europe.

DETAILED DESCRIPTION:
Synthetic ACTH (Synacthen Depot) has been used in the treatment of Nephrotic Syndrome in Europe. It has been proven effective in treating idiopathic membranous nephropathy and other various diagnoses involving the kidneys. However, Synacthen is not available in the United States. The only preparation available is the H.P. Acthar Gel (repository corticotrophin) which has been widely used in the treatment of infantile spasms and has been available longer than Synacthen. Therefore, we are conducting this study to determine if H.P. Acthar Gel (repository corticotrophin) is as effective in reducing protein in the urine as seen in synthetic ACTH in Europe.

ELIGIBILITY:
Inclusion Criteria:

* Nephrotic Syndrome with a minimal of 3.5grams of protein per 24 hr period, measured via either 24hr urine collection or spot protein to creatinine ratio.
* Males and post-menopausal, surgically sterile, or non-lactating and non-pregnant females using adequate contraception
* Biopsy proven diagnosis of nephrotic syndrome due to Lupus glomerulonephritis, Membranous nephropathy, Focal segmental glomerulosclerosis, Minimal Change disease, Diabetic nephropathy (type 2)or IgA nephropathy.
* Greater than 18 years of age
* Willing and able to give informed consent
* Diabetics are on insulin or willing to start insulin during the study

Exclusion Criteria:

* Previous intolerance to native ACTH or proteins of porcine origin
* History of scleroderma, osteoporosis, systemic fungal infections, ocular herpes simplex, recent surgery, history of or the presence of peptic ulcer, primary adrenocortical insufficiency or adrenocortical hyperfunction.
* Expected to begin renal replacement therapy or receive a transplant within the next year.
* Recent cardiovascular event within 3 months of screening including: Myocardial Infarction, CVA, TIA, New York Heart Association Functional Class III or IV failure, Obstructive valvular heart disease, or hypertrophic cardiomyopathy, second or third degree atrioventricular block not successfully treated with a pacemaker.
* History of HIV
* Know peptic ulcer disease.
* SBP> 160 or DBP > 100 at time of enrollment
* New diagnosis of cancer or recurrent cancer within 2 years of screening
* History of alcohol or drug abuse within 12 months of study entry.
* Receipt of any investigational drug within 30 days of enrollment.
* Anticipated major surgery during trial period
* Psychiatric disorder that interferes with the patient's ability to comply with the protocol.
* Inability to cooperate with study personnel or history of noncompliance to medical management
* Active infection within 1 month of screening
* Poorly controlled diabetes with an HbA1C > 10%
* Type 1 diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Acthar has the same anti-proteinuric effects in a wide range of glomerulonephropaties as seen with synthetic ACTH (Synacthen) in Europe | 6 months

SECONDARY OUTCOMES:
Acthar has similar anti-lipid effects as seen with Synacthen. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sungchun Lee, M.D., Principal Investigator — Arizona Kidney Disease and Hypertension Center
Locations (1):
- AKDHC, Phoenix, Arizona, United States